CLINICAL TRIAL: NCT01984866
Title: Complete Pathological Response Prediction After Neoadjuvant Treatment Using Excisional Biopsy By Radiofrequency In Breast Cancer From II-III UICC Stages.
Brief Title: CPR Prediction After Neoadjuvant Using Excisional Biopsy By Radiofrequency In Breast Cancer From II-III UICC Stages.
Status: Terminated | Type: Observational
Why Stopped: Recruitment was very low.
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Responsible Party: Sponsor
Other Study IDs: GOMHGUGM032012
Record Dates: First submitted 2013-10-10; First posted 2013-11-15 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Triple Negative, HER2+, Luminal B Breast Tumors (Stages II-III)in Female Patients
Keywords: CPR: Complete Pathological Response

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tissue samples from breast tumors

GROUPS / COHORTS (1):
- Breast tumors sensitive to neoadjuvant: Treated patients as usual clinical practice with unicentered tumors in stages II or III and good response determined by MR after 6 cycles of treatment (less than 2 cm apparent residual injury) will be consecutively subjected to radiofrequency biopsy and the surgery previously established for each case (Tumorectomy or mastectomy). Before surgery, the sentinel node will be biopsied in order to define the surgical treatment on the axilla (none in case of negative sentinel node, axillary lymphadenectomy if positive).
  The tumor samples obtained by percutaneous radiofrequency and mastectomy-Tumorectomy biopsy will be studied thoroughly to define the correlation between the two.

SUMMARY:
This project aims to determine whether biopsy using radiofrequency is a procedure suitable for this patient selection. Findings from biopsy will be correlated with the conventional surgery ones. If the technique is validated to predict the presence or absence of residual tumor, breast surgery could be avoided in cases of absence of tumor.

DETAILED DESCRIPTION:
Breast cancer is a set of at least 4 different diseases, currently known as intrinsic genomic subtypes. Two of them are the so-called HER2-enriched, characterized by the HER-2 oncogene amplification, and the basal-like, which correlates closely with some of the triple negative tumors (TNBC). These subtypes are very sensitive to the primary medical treatment (neoadjuvant or Presurgical). The use of modern medical treatments as initial treatment, can allow the complete disappearance of cancer in the breast and axilla (pathologic complete response, CPR) in 40% of patients with TNBC and around 60% of patients with HER2-positive tumors in stage II and III.

The need of local surgery in patients where the tumor disappeared completely (CPR) after primary medical treatment, is recently questioned, the improvement is not clear and radiotherapy could be sufficient to assure the locoregional disease control.

The use of conventional diagnostic techniques (MRI, ultrasound, mammography and PET) is not enough reliable to determine the pathological complete response, making difficult to adopt an attitude of surgical abstention. The existence of a minimally invasive technique that could reliably determine the absence of cancer after primary medical treatment surgery, could avoid the surgery in these cases.

Percutaneous biopsy guided by ultrasound radiofrequency is a technique that allows the complete resection of breast lesions up to 2 cm of diameter with minimal aggression to the mammary gland from the area of the initial tumor after the neoadjuvant treatment.

Several studies report the use of this technique in patients with breast cancer. Results show a good tolerability of the technique by the patients and suggest that it would not only reduce the need of the re-excision, but also reduce the rate of local recurrence due to radiation absence.

Biopsy using radiofrequency could be useful to confirm CPR in patients with triple-negative and HER2-positive tumors and several luminal B tumors and good response previously determined by conventional methods (MR in particular). Despite that, new prospective studies to analyse the reliability in patients selection with CPR and could avoid the traditional surgery are needed.

To confirm this hypothesis, a group of 100 treated patients with unicentered tumors in stages II or III and good response determined by MR after 6 cycles of treatment (less than 2 cm apparent residual injury) will be consecutively subjected to radiofrequency biopsy and the surgery previously established for each case (Tumorectomy or mastectomy). Before surgery, the sentinel node will be biopsied in order to define the surgical treatment on the axilla (none in case of negative sentinel node, axillary lymphadenectomy if positive).

The tumor samples obtained by percutaneous radiofrequency and mastectomy-Tumorectomy biopsy will be studied thoroughly to define the correlation between the two.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent Form signed
* Adequate Performance status (ECOG 0-1)
* Female patients with unifocal breast tumors (stages II-III, TN, HER2+ or Luminal B) very sensitive to neoadjuvant medical treatment (5 to 6 months in accordance with the current standard)
* Patients who submit clinical-radiologic greater response to the treatment administered (equal to or less than 1.5 cm in NMR residual tumor)

Exclusion Criteria:

* Ki67<14%
* Excisional biopsy Contraindications

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients with breast tumors sensitive to neoadjuvancy
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-07; Primary Completion 2018-04 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
determination of the negative predictive value (NPV) of the excisional biopsy technique | up to 15 months
  Proportion of biopsies which PCR, are really PCR in the surgical specimen.

SECONDARY OUTCOMES:
Evaluation of sensitivity and specificity of the excisional biopsy by radiofrequency technique | up to 15 months
  * Determine the sensitivity and specificity of excisional biopsy, radiofrequency technique, to classify correctly the stage of the tumor in the breast after neoadjuvant therapy.
  * Determine the positive predictive value (proportion of biopsies which are not CPR and actually have tumor in the surgical specimen).
  * Describe the side effects of the excisional biopsy technique by radiofrequency.
  * Describe the technical problems associated to excisional biopsy technique by radiofrequency.
  * Assess the concordance between the responses obtained in breast MRI and the previous reported in the anatomy-pathological study.
  * Determine the % of cases in which surgery could have been avoided within the group defined in the study.
  * Estimate the economic cost of excisional biopsy with standard therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital General Universitario Gregorio Marañón, Madrid, Spain